CLINICAL TRIAL: NCT04248413
Title: Blood Flow Restriction Training Following Acute Shoulder Injury In Baseball Players: Assessment of Efficacy in Return to Sport
Brief Title: Return to Baseball After BFR Therapy for Shoulder Injury
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Too many obstacles starting study
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00062859
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Musculoskeletal Injury
Keywords: Shoulder injury; Baseball injury; Muscle strength
MeSH Terms: conditions — Shoulder Injuries | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: The purpose of the study is to 1) evaluate patient reported outcomes and return to play in baseball athletes undergoing rehabilitation with blood flow restriction (BFR) therapy for shoulder injury and 2) evaluate changes in blood biomarkers to assess the mechanism of action of BFR therapy in injured athletes.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The PI who will be performing the analysis will be blinded to patients who underwent routine physical rehabilitation vs those who underwent routine rehabilitation plus blood flow restriction therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard rehabilitation protocol (Other): Patients with non-operative rotator cuff and biceps tendinopathy assigned to this study arm will undergo the standardized physical rehabilitation protocol at our institution.
  Interventions: Other: Standard physical rehabilitation
- Standard rehabilitation plus Blood Flow Restriction Therapy (Experimental): Patients with non-operative rotator cuff and biceps tendinopathy assigned to this study arm will undergo the standardized physical rehabilitation protocol at our institution in addition to the BFR therapy. Per recommendations of Owens Recovery Science, the organization responsible for certifying physical therapists in BFR therapy, the therapy will take place concurrently throughout the duration of the rehabilitation.
  Interventions: Device: Blood Flow Restriction Therapy; Other: Standard physical rehabilitation

INTERVENTIONS:
Device: Blood Flow Restriction Therapy — The blood flow restriction cuff, which is regulated by the FDA under 878.5910 and is registered under number 9681444, is manufactured by Delfi Medical. The cuff will be used as recommended by the manufacturer and Owens Recovery Science, the company who provides certificating of blood flow restriction training.
  Arms: Standard rehabilitation plus Blood Flow Restriction Therapy
Other: Standard physical rehabilitation — Patients diagnosed with non-operative rotator cuff or biceps tendinopathy will undergo physical rehabilitation under the supervision of the same physical therapists who will be performing the BFR therapy.

SUMMARY:
The literature is limited on whether BFR therapy provides improved return to function after acute rotator cuff or biceps rehabilitation in non-operative cases, and whether there is a clear mechanism of action in musculotendinous repair after BFR therapy. The purpose of the study is to 1) evaluate patient reported outcomes and return to play in baseball athletes undergoing rehabilitation with blood flow restriction (BFR) therapy for shoulder injury and 2) evaluate changes in blood biomarkers to assess the mechanism of action of BFR therapy in injured athletes. Investigators will perform a randomized blinded placebo-controlled trial of 2 separate study populations: 1) baseball players with biceps or rotator cuff tendinopathy undergoing non-operative treatment with BFR therapy incorporated into routine physical rehabilitation and 2) baseball players with biceps or rotator cuff tendinopathy undergoing non-operative treatment with routine physical rehabilitation alone.

Primary outcomes will be functional outcomes and evaluation of return to sport. Functional outcomes will be evaluated using validated patient reported outcome surveys that are upper extremity-specific. Return to sport will be assessed by evaluating time to receiving clearance for returning to routine practices and reported level of physical performance and re-injury. Secondary outcomes will be measurement in muscle strength and blood biomarkers, as well as evaluation of 3D throwing motion. Strength will be measured using a biodex system at baseline prior to beginning physical rehabilitation, half-way through the rehabilitation protocol +/- BFR phase, and once cleared for return to play. Blood biomarkers GH, IGF-I, and IL-6 will be quantified at the same time points in order to investigate the mechanism of action of BFR on tissue repair. Patients will be followed longitudinally during this time for rates of reinjury.

DETAILED DESCRIPTION:
This study will evaluate the efficacy of BFR therapy in physical rehabilitation for baseball athletes with non-operative biceps or rotator cuff tendinopathy. This will be directly measured by evaluation of upper extremity biomechanics measurements, strength testing, patient reported functional outcome scores, and identifying time required for clearance of return to sport. These outcomes in patients undergoing BFR therapy in addition to traditional rehabilitation will be compared to patients undergoing traditional rehabilitation only.

ELIGIBILITY:
Inclusion Criteria:

* any injured baseball athletes ages 14 to 25 years with clinical and radiographic examination (MRI) consistent with a formal diagnosis of non-operative rotator cuff and/or biceps tendinopathy
* no prior upper extremity ipsilateral procedures or history of deep vein thrombosis

Exclusion Criteria:

* patients younger than 14 or older than 25 years of age
* non-native English speakers
* a history of revision surgery or prior ipsilateral upper extremity surgery, concomitant ligamentous, tendinous, or cartilage injury that would alter postoperative rehabilitation protocol
* inability to comply with the proposed follow-up clinic visits
* patients lacking decisional capacity.

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) questionnaire | Questionnaire assigned at baseline prior to the rehabilitation protocol.
  Patient-reported outcome questionnaire with a score ranging from 0 to 100. A higher score denotes a better outcome.
American Shoulder and Elbow Surgeons (ASES) questionnaire | Questionnaire assigned at the half-way point during the rehabilitation protocol, which is approximately 6-7 weeks from start of rehabilitation.
  Patient-reported outcome questionnaire with a score ranging from 0 to 100. A higher score denotes a better outcome.
American Shoulder and Elbow Surgeons (ASES) questionnaire | Questionnaire assigned at the end of the rehabilitation protocol, corresponding to when the patient is cleared to return to sport, which is approximately 12-14 weeks from start of rehabilitation.
  Patient-reported outcome questionnaire with a score ranging from 0 to 100. A higher score denotes a better outcome.
American Shoulder and Elbow Surgeons (ASES) questionnaire | Questionnaire assigned 6-months after completing the rehabilitation protocol.
  Patient-reported outcome questionnaire with a score ranging from 0 to 100. A higher score denotes a better outcome.
American Shoulder and Elbow Surgeons (ASES) questionnaire | Questionnaire assigned 12-months after completing the rehabilitation protocol.
  Patient-reported outcome questionnaire with a score ranging from 0 to 100. A higher score denotes a better outcome.
Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire | Questionnaire assigned at baseline prior to the rehabilitation protocol.
  Patient-reported outcome questionnaire with a score ranging from 0 to 100. A lower score denotes a better outcome.
Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire | Questionnaire assigned at the half-way point during the rehabilitation protocol, which is approximately 6-7 weeks from start of rehabilitation.
  Patient-reported outcome questionnaire with a score ranging from 0 to 100. A lower score denotes a better outcome.
Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire | Questionnaire assigned at the end of the rehabilitation protocol, corresponding to when the patient is cleared to return to sport, which is approximately 12-14 weeks from start of rehabilitation.
  Patient-reported outcome questionnaire with a score ranging from 0 to 100. A lower score denotes a better outcome.
Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire | Questionnaire assigned 6-months after completing the rehabilitation protocol.
  Patient-reported outcome questionnaire with a score ranging from 0 to 100. A lower score denotes a better outcome.
Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire | Questionnaire assigned 12-months after completing the rehabilitation protocol.
  Patient-reported outcome questionnaire with a score ranging from 0 to 100. A lower score denotes a better outcome.
Return to sport questionnaire | Questionnaire assigned 6-months after completing the rehabilitation protocol.
  Patient-reported questionnaire evaluating physical performance and re-injury after undergoing rehabilitation. Patient-reported outcome questionnaire with a score ranging from 0 to 10. A higher score denotes a better outcome.
Return to sport questionnaire | Questionnaire assigned 12-months after completing the rehabilitation protocol.
  Patient-reported questionnaire evaluating physical performance and re-injury after undergoing rehabilitation. Patient-reported outcome questionnaire with a score ranging from 0 to 10. A higher score denotes a better outcome.

SECONDARY OUTCOMES:
Muscle Strength | Measured at baseline prior to the rehabilitation protocol.
  Upper extremity muscle strength will be measured using a biodex strength training machine. Physiological parameters will include peak torque (measured as Newtons) and time to peak torque (measured in seconds), which is time from the start of the muscular contraction to the point of highest torque.
Muscle Strength | Measured at the half-way point during the rehabilitation protocol, which is approximately 6-7 weeks from start of rehabilitation.
  Upper extremity muscle strength will be measured using a biodex strength training machine. Physiological parameters will include peak torque (measured as Newtons) and time to peak torque (measured in seconds), which is time from the start of the muscular contraction to the point of highest torque.
Muscle Strength | Measured at the end of the rehabilitation protocol, corresponding to when the patient is cleared to return to sport, which is approximately 12-14 weeks from start of rehabilitation.
  Upper extremity muscle strength will be measured using a biodex strength training machine. Physiological parameters will include peak torque (measured as Newtons) and time to peak torque (measured in seconds), which is time from the start of the muscular contraction to the point of highest torque.
3D throwing motion analysis | Performed at baseline prior to the rehabilitation protocol.
  Throwing biomechanics will be evaluated using 3D motion analysis.
3D throwing motion analysis | Performed at the end of the rehabilitation protocol, corresponding to when the patient is cleared to return to sport, which is approximately 12-14 weeks from start of rehabilitation.
  Throwing biomechanics will be evaluated using 3D motion analysis and will be compared to 3D throwing motion captured at baseline prior to beginning rehabilitation.
Human Growth Hormone (GH) | Measured at baseline prior to the rehabilitation protocol.
  GH will be quantified from blood draws and compared between the two study groups.
Human Growth Hormone (GH) | Measured at the half-way point during the rehabilitation protocol, which is approximately 6-7 weeks from start of rehabilitation.
  GH will be quantified from blood draws and compared between the two study groups.
Human Growth Hormone (GH) | Measured at the end of the rehabilitation protocol, corresponding to when the patient is cleared to return to sport, which is approximately 12-14 weeks from start of rehabilitation.
  GH will be quantified from blood draws and compared between the two study groups.
Interleukin 6 (IL-6) | Measured at baseline prior to the rehabilitation protocol.
  IL-6 will be quantified from blood draws and compared between the two study groups.
Interleukin 6 (IL-6) | Measured at the half-way point during the rehabilitation protocol, which is approximately 6-7 weeks from start of rehabilitation.
  IL-6 will be quantified from blood draws and compared between the two study groups.
Interleukin 6 (IL-6) | Measured at the end of the rehabilitation protocol, corresponding to when the patient is cleared to return to sport, which is approximately 12-14 weeks from start of rehabilitation.
  IL-6 will be quantified from blood draws and compared between the two study groups.
Insulin-Like Growth Factor (IGF) | Measured at baseline prior to the rehabilitation protocol.
  IGF will be quantified from blood draws and compared between the two study groups.
Insulin-Like Growth Factor (IGF) | Measured at the half-way point during the rehabilitation protocol, which is approximately 6-7 weeks from start of rehabilitation.
  IGF will be quantified from blood draws and compared between the two study groups.
Insulin-Like Growth Factor (IGF) | Measured at the end of the rehabilitation protocol, corresponding to when the patient is cleared to return to sport, which is approximately 12-14 weeks from start of rehabilitation.
  IGF will be quantified from blood draws and compared between the two study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen F Nicholson, PhD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abe T, Fujita S, Nakajima T, Sakamaki M, Ozaki H, Ogasawara R, Sugaya M, Kudo M, Kurano M, Yasuda T, Sato Y, Ohshima H, Mukai C, Ishii N. Effects of Low-Intensity Cycle Training with Restricted Leg Blood Flow on Thigh Muscle Volume and VO2MAX in Young Men. J Sports Sci Med. 2010 Sep 1;9(3):452-8. eCollection 2010. PMID 24149640
- [Background] Abe T, Yasuda T, Midorikawa T, et al. Skeletal muscle size and circulating IGF-1 are increased after two weeks of twice daily "KAATSU" resistance training. International Journal of KAATSU Training Research. 2005;1(1):6-12.
- [Background] Blair JA, Eisenstein ED, Pierrie SN, Gordon W, Owens JG, Hsu JR. Lower Extremity Limb Salvage: Lessons Learned From 14 Years at War. J Orthop Trauma. 2016 Oct;30 Suppl 3:S11-S15. doi: 10.1097/BOT.0000000000000669. PMID 27661420
- [Background] Bowman EN, Elshaar R, Milligan H, Jue G, Mohr K, Brown P, Watanabe DM, Limpisvasti O. Proximal, Distal, and Contralateral Effects of Blood Flow Restriction Training on the Lower Extremities: A Randomized Controlled Trial. Sports Health. 2019 Mar/Apr;11(2):149-156. doi: 10.1177/1941738118821929. Epub 2019 Jan 14. PMID 30638439
- [Background] Burkhart SS, Morgan CD, Kibler WB. The disabled throwing shoulder: spectrum of pathology Part I: pathoanatomy and biomechanics. Arthroscopy. 2003 Apr;19(4):404-20. doi: 10.1053/jars.2003.50128. PMID 12671624
- [Background] Cancio J, Rhee P. Blood Flow Restriction Therapy after Non-Operative Management of Distal Radius Fracture: A Randomized Controlled Pilot Study. Journal of Hand Therapy. 2018;31(1).
- [Background] Clarsen B, Myklebust G, Bahr R. Development and validation of a new method for the registration of overuse injuries in sports injury epidemiology: the Oslo Sports Trauma Research Centre (OSTRC) overuse injury questionnaire. Br J Sports Med. 2013 May;47(8):495-502. doi: 10.1136/bjsports-2012-091524. Epub 2012 Oct 4. PMID 23038786
- [Background] Conte S, Camp CL, Dines JS. Injury Trends in Major League Baseball Over 18 Seasons: 1998-2015. Am J Orthop (Belle Mead NJ). 2016 Mar-Apr;45(3):116-23. PMID 26991562
- [Background] Credeur DP, Hollis BC, Welsch MA. Effects of handgrip training with venous restriction on brachial artery vasodilation. Med Sci Sports Exerc. 2010 Jul;42(7):1296-302. doi: 10.1249/MSS.0b013e3181ca7b06. PMID 20019641
- [Background] Cvetanovich GL, Gowd AK, Liu JN, Nwachukwu BU, Cabarcas BC, Cole BJ, Forsythe B, Romeo AA, Verma NN. Establishing clinically significant outcome after arthroscopic rotator cuff repair. J Shoulder Elbow Surg. 2019 May;28(5):939-948. doi: 10.1016/j.jse.2018.10.013. Epub 2019 Jan 24. PMID 30685283
- [Background] Dahlgren LA, Mohammed HO, Nixon AJ. Temporal expression of growth factors and matrix molecules in healing tendon lesions. J Orthop Res. 2005 Jan;23(1):84-92. doi: 10.1016/j.orthres.2004.05.007. PMID 15607879
- [Background] Dankel SJ, Jessee MB, Abe T, Loenneke JP. The Effects of Blood Flow Restriction on Upper-Body Musculature Located Distal and Proximal to Applied Pressure. Sports Med. 2016 Jan;46(1):23-33. doi: 10.1007/s40279-015-0407-7. PMID 26446893
- [Background] Dines JS, Frank JB, Akerman M, Yocum LA. Glenohumeral internal rotation deficits in baseball players with ulnar collateral ligament insufficiency. Am J Sports Med. 2009 Mar;37(3):566-70. doi: 10.1177/0363546508326712. Epub 2008 Dec 4. PMID 19059890
- [Background] Erickson LN, Lucas KCH, Davis KA, Jacobs CA, Thompson KL, Hardy PA, Andersen AH, Fry CS, Noehren BW. Effect of Blood Flow Restriction Training on Quadriceps Muscle Strength, Morphology, Physiology, and Knee Biomechanics Before and After Anterior Cruciate Ligament Reconstruction: Protocol for a Randomized Clinical Trial. Phys Ther. 2019 Aug 1;99(8):1010-1019. doi: 10.1093/ptj/pzz062. PMID 30951598
- [Background] Escamilla RF, Barrentine SW, Fleisig GS, Zheng N, Takada Y, Kingsley D, Andrews JR. Pitching biomechanics as a pitcher approaches muscular fatigue during a simulated baseball game. Am J Sports Med. 2007 Jan;35(1):23-33. doi: 10.1177/0363546506293025. Epub 2006 Sep 14. PMID 16973902
- [Background] Fleisig GS, Barrentine SW, Zheng N, Escamilla RF, Andrews JR. Kinematic and kinetic comparison of baseball pitching among various levels of development. J Biomech. 1999 Dec;32(12):1371-5. doi: 10.1016/s0021-9290(99)00127-x. PMID 10569718
- [Background] Fujita S, Abe T, Drummond MJ, Cadenas JG, Dreyer HC, Sato Y, Volpi E, Rasmussen BB. Blood flow restriction during low-intensity resistance exercise increases S6K1 phosphorylation and muscle protein synthesis. J Appl Physiol (1985). 2007 Sep;103(3):903-10. doi: 10.1152/japplphysiol.00195.2007. Epub 2007 Jun 14. PMID 17569770
- [Background] Gao S, Durstine JL, Koh HJ, Carver WE, Frizzell N, Carson JA. Acute myotube protein synthesis regulation by IL-6-related cytokines. Am J Physiol Cell Physiol. 2017 Nov 1;313(5):C487-C500. doi: 10.1152/ajpcell.00112.2017. Epub 2017 Aug 2. PMID 28768641
- [Background] Garrison JC, Johnston C, Conway JE. BASEBALL PLAYERS WITH ULNAR COLLATERAL LIGAMENT TEARS DEMONSTRATE DECREASED ROTATOR CUFF STRENGTH COMPARED TO HEALTHY CONTROLS. Int J Sports Phys Ther. 2015 Aug;10(4):476-81. PMID 26346550
- [Background] Gilliam BD, Douglas L, Fleisig GS, Aune KT, Mason KA, Dugas JR, Cain EL Jr, Ostrander RV, Andrews JR. Return to Play and Outcomes in Baseball Players After Superior Labral Anterior-Posterior Repairs. Am J Sports Med. 2018 Jan;46(1):109-115. doi: 10.1177/0363546517728256. Epub 2017 Sep 25. PMID 28942657
- [Background] Goto K, Ishii N, Kizuka T, Takamatsu K. The impact of metabolic stress on hormonal responses and muscular adaptations. Med Sci Sports Exerc. 2005 Jun;37(6):955-63. PMID 15947720
- [Background] Hylden C, Burns T, Stinner D, Owens J. Blood flow restriction rehabilitation for extremity weakness: a case series. J Spec Oper Med. 2015 Spring;15(1):50-6. PMID 25770798
- [Background] Iversen E, Rostad V, Larmo A. Intermittent blood flow restriction does not reduce atrophy following anterior cruciate ligament reconstruction. J Sport Health Sci. 2016 Mar;5(1):115-118. doi: 10.1016/j.jshs.2014.12.005. Epub 2015 Apr 18. PMID 30356481
- [Background] Jo CH, Park JW, Shin JS. Changes of Muscle Atrophy According to the Immediate Postoperative Time Point in Magnetic Resonance Imaging After Arthroscopic Rotator Cuff Repair. Arthroscopy. 2016 Dec;32(12):2477-2487. doi: 10.1016/j.arthro.2016.04.032. Epub 2016 Jun 22. PMID 27344233
- [Background] Jobe FW, Kvitne RS, Giangarra CE. Shoulder pain in the overhand or throwing athlete. The relationship of anterior instability and rotator cuff impingement. Orthop Rev. 1989 Sep;18(9):963-75. PMID 2797861
- [Background] Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics. 2005;4(4):287-291.
- [Background] Ladlow P, Coppack RJ, Dharm-Datta S, Conway D, Sellon E, Patterson SD, Bennett AN. Low-Load Resistance Training With Blood Flow Restriction Improves Clinical Outcomes in Musculoskeletal Rehabilitation: A Single-Blind Randomized Controlled Trial. Front Physiol. 2018 Sep 10;9:1269. doi: 10.3389/fphys.2018.01269. eCollection 2018. PMID 30246795
- [Background] Laurentino GC, Ugrinowitsch C, Roschel H, Aoki MS, Soares AG, Neves M Jr, Aihara AY, Fernandes Ada R, Tricoli V. Strength training with blood flow restriction diminishes myostatin gene expression. Med Sci Sports Exerc. 2012 Mar;44(3):406-12. doi: 10.1249/MSS.0b013e318233b4bc. PMID 21900845
- [Background] Loenneke JP, Thiebaud RS, Abe T, Bemben MG. Blood flow restriction pressure recommendations: the hormesis hypothesis. Med Hypotheses. 2014 May;82(5):623-6. doi: 10.1016/j.mehy.2014.02.023. Epub 2014 Mar 2. PMID 24636784
- [Background] Makhni EC, Higgins JD, Hamamoto JT, Cole BJ, Romeo AA, Verma NN. Patient Compliance With Electronic Patient Reported Outcomes Following Shoulder Arthroscopy. Arthroscopy. 2017 Nov;33(11):1940-1946. doi: 10.1016/j.arthro.2017.06.016. Epub 2017 Sep 27. PMID 28958797
- [Background] Manini TM, Yarrow JF, Buford TW, Clark BC, Conover CF, Borst SE. Growth hormone responses to acute resistance exercise with vascular restriction in young and old men. Growth Horm IGF Res. 2012 Oct;22(5):167-72. doi: 10.1016/j.ghir.2012.05.002. Epub 2012 Jun 23. PMID 22727808
- [Background] Manske R, Prohaska D. Superior labrum anterior to posterior (SLAP) rehabilitation in the overhead athlete. Phys Ther Sport. 2010 Nov;11(4):110-21. doi: 10.1016/j.ptsp.2010.06.004. Epub 2010 Jul 27. PMID 21055704
- [Background] Mascarenhas R, Verma NN. Editorial Commentary: Muscle Atrophy After Arthroscopic Rotator Cuff Repair-Reversible? Arthroscopy. 2016 Dec;32(12):2488-2489. doi: 10.1016/j.arthro.2016.08.007. PMID 27916184
- [Background] McLeod WD, Andrews JR. Mechanisms of shoulder injuries. Phys Ther. 1986 Dec;66(12):1901-4. doi: 10.1093/ptj/66.12.1901. PMID 3786420
- [Background] Meister K, Day T, Horodyski M, Kaminski TW, Wasik MP, Tillman S. Rotational motion changes in the glenohumeral joint of the adolescent/Little League baseball player. Am J Sports Med. 2005 May;33(5):693-8. doi: 10.1177/0363546504269936. Epub 2005 Feb 16. PMID 15722284
- [Background] Moore DR, Burgomaster KA, Schofield LM, Gibala MJ, Sale DG, Phillips SM. Neuromuscular adaptations in human muscle following low intensity resistance training with vascular occlusion. Eur J Appl Physiol. 2004 Aug;92(4-5):399-406. doi: 10.1007/s00421-004-1072-y. PMID 15205956
- [Background] Myers JB, Laudner KG, Pasquale MR, Bradley JP, Lephart SM. Glenohumeral range of motion deficits and posterior shoulder tightness in throwers with pathologic internal impingement. Am J Sports Med. 2006 Mar;34(3):385-91. doi: 10.1177/0363546505281804. Epub 2005 Nov 22. PMID 16303877
- [Background] Ohta H, Kurosawa H, Ikeda H, Iwase Y, Satou N, Nakamura S. Low-load resistance muscular training with moderate restriction of blood flow after anterior cruciate ligament reconstruction. Acta Orthop Scand. 2003 Feb;74(1):62-8. doi: 10.1080/00016470310013680. PMID 12635796
- [Background] Olesen JL, Heinemeier KM, Gemmer C, Kjaer M, Flyvbjerg A, Langberg H. Exercise-dependent IGF-I, IGFBPs, and type I collagen changes in human peritendinous connective tissue determined by microdialysis. J Appl Physiol (1985). 2007 Jan;102(1):214-20. doi: 10.1152/japplphysiol.01205.2005. Epub 2006 Sep 14. PMID 16973813
- [Background] Oyama S. Baseball pitching kinematics, joint loads, and injury prevention. Journal of Sport and Health Science. 2012;1(2):80-91.
- [Background] Patterson SD, Ferguson RA. Increase in calf post-occlusive blood flow and strength following short-term resistance exercise training with blood flow restriction in young women. Eur J Appl Physiol. 2010 Mar;108(5):1025-33. doi: 10.1007/s00421-009-1309-x. Epub 2009 Dec 11. PMID 20012448
- [Background] Posner M, Cameron KL, Wolf JM, Belmont PJ Jr, Owens BD. Epidemiology of Major League Baseball injuries. Am J Sports Med. 2011 Aug;39(8):1676-80. doi: 10.1177/0363546511411700. Epub 2011 Jun 27. PMID 21709023
- [Background] Poton R, Polito MD. Hemodynamic response to resistance exercise with and without blood flow restriction in healthy subjects. Clin Physiol Funct Imaging. 2016 May;36(3):231-6. doi: 10.1111/cpf.12218. Epub 2014 Nov 27. PMID 25431280
- [Background] Reeves GV, Kraemer RR, Hollander DB, Clavier J, Thomas C, Francois M, Castracane VD. Comparison of hormone responses following light resistance exercise with partial vascular occlusion and moderately difficult resistance exercise without occlusion. J Appl Physiol (1985). 2006 Dec;101(6):1616-22. doi: 10.1152/japplphysiol.00440.2006. Epub 2006 Aug 10. PMID 16902061
- [Background] Rossi FE, de Freitas MC, Zanchi NE, Lira FS, Cholewa JM. The Role of Inflammation and Immune Cells in Blood Flow Restriction Training Adaptation: A Review. Front Physiol. 2018 Oct 9;9:1376. doi: 10.3389/fphys.2018.01376. eCollection 2018. PMID 30356748
- [Background] Ruotolo C, Price E, Panchal A. Loss of total arc of motion in collegiate baseball players. J Shoulder Elbow Surg. 2006 Jan-Feb;15(1):67-71. doi: 10.1016/j.jse.2005.05.006. PMID 16414471
- [Background] Sciore P, Boykiw R, Hart DA. Semiquantitative reverse transcription-polymerase chain reaction analysis of mRNA for growth factors and growth factor receptors from normal and healing rabbit medial collateral ligament tissue. J Orthop Res. 1998 Jul;16(4):429-37. doi: 10.1002/jor.1100160406. PMID 9747783
- [Background] Serrano AL, Baeza-Raja B, Perdiguero E, Jardi M, Munoz-Canoves P. Interleukin-6 is an essential regulator of satellite cell-mediated skeletal muscle hypertrophy. Cell Metab. 2008 Jan;7(1):33-44. doi: 10.1016/j.cmet.2007.11.011. PMID 18177723
- [Background] Shimizu R, Hotta K, Yamamoto S, Matsumoto T, Kamiya K, Kato M, Hamazaki N, Kamekawa D, Akiyama A, Kamada Y, Tanaka S, Masuda T. Low-intensity resistance training with blood flow restriction improves vascular endothelial function and peripheral blood circulation in healthy elderly people. Eur J Appl Physiol. 2016 Apr;116(4):749-57. doi: 10.1007/s00421-016-3328-8. Epub 2016 Jan 28. PMID 26822582
- [Background] Steinberg L. Baseball Has A Serious Injury Problem. Forbes. Available at: https://www.forbes.com/sites/leighsteinberg/2018/07/24/baseball-the-most-dangerous-sport-in-america/. Accessed November 2, 2018.
- [Background] Takano H, Morita T, Iida H, Asada K, Kato M, Uno K, Hirose K, Matsumoto A, Takenaka K, Hirata Y, Eto F, Nagai R, Sato Y, Nakajima T. Hemodynamic and hormonal responses to a short-term low-intensity resistance exercise with the reduction of muscle blood flow. Eur J Appl Physiol. 2005 Sep;95(1):65-73. doi: 10.1007/s00421-005-1389-1. Epub 2005 Jun 15. PMID 15959798
- [Background] Takarada Y, Nakamura Y, Aruga S, Onda T, Miyazaki S, Ishii N. Rapid increase in plasma growth hormone after low-intensity resistance exercise with vascular occlusion. J Appl Physiol (1985). 2000 Jan;88(1):61-5. doi: 10.1152/jappl.2000.88.1.61. PMID 10642363
- [Background] Takarada Y, Takazawa H, Ishii N. Applications of vascular occlusion diminish disuse atrophy of knee extensor muscles. Med Sci Sports Exerc. 2000 Dec;32(12):2035-9. doi: 10.1097/00005768-200012000-00011. PMID 11128848
- [Background] Tennent DJ, Burns TC, Johnson AE, Owens JG, Hylden CM. Blood Flow Restriction Training for Postoperative Lower-Extremity Weakness: A Report of Three Cases. Curr Sports Med Rep. 2018 Apr;17(4):119-122. doi: 10.1249/JSR.0000000000000470. No abstract available. PMID 29629970
- [Background] Tennent DJ, Hylden CM, Johnson AE, Burns TC, Wilken JM, Owens JG. Blood Flow Restriction Training After Knee Arthroscopy: A Randomized Controlled Pilot Study. Clin J Sport Med. 2017 May;27(3):245-252. doi: 10.1097/JSM.0000000000000377. PMID 27749358
- [Background] Walch G, Boileau P, Noel E, Donell ST. Impingement of the deep surface of the supraspinatus tendon on the posterosuperior glenoid rim: An arthroscopic study. J Shoulder Elbow Surg. 1992 Sep;1(5):238-45. doi: 10.1016/S1058-2746(09)80065-7. Epub 2009 Feb 19. PMID 22959196
- [Background] Wall BT, Dirks ML, Snijders T, Senden JM, Dolmans J, van Loon LJ. Substantial skeletal muscle loss occurs during only 5 days of disuse. Acta Physiol (Oxf). 2014 Mar;210(3):600-11. doi: 10.1111/apha.12190. Epub 2013 Dec 5. PMID 24168489
- [Background] Werner SL, Gill TJ, Murray TA, Cook TD, Hawkins RJ. Relationships between throwing mechanics and shoulder distraction in professional baseball pitchers. Am J Sports Med. 2001 May-Jun;29(3):354-8. doi: 10.1177/03635465010290031701. PMID 11394608
- [Background] Werner SL, Guido JA Jr, Stewart GW, McNeice RP, VanDyke T, Jones DG. Relationships between throwing mechanics and shoulder distraction in collegiate baseball pitchers. J Shoulder Elbow Surg. 2007 Jan-Feb;16(1):37-42. doi: 10.1016/j.jse.2006.05.007. Epub 2006 Dec 12. PMID 17169584
- [Background] Wilk KE, Macrina LC, Fleisig GS, Aune KT, Porterfield RA, Harker P, Evans TJ, Andrews JR. Deficits in glenohumeral passive range of motion increase risk of elbow injury in professional baseball pitchers: a prospective study. Am J Sports Med. 2014 Sep;42(9):2075-81. doi: 10.1177/0363546514538391. Epub 2014 Jun 18. PMID 24944295
- [Background] Yasuda T, Loenneke JP, Thiebaud RS, Abe T. Effects of blood flow restricted low-intensity concentric or eccentric training on muscle size and strength. PLoS One. 2012;7(12):e52843. doi: 10.1371/journal.pone.0052843. Epub 2012 Dec 31. PMID 23300795
- [Background] Yoon MS. mTOR as a Key Regulator in Maintaining Skeletal Muscle Mass. Front Physiol. 2017 Oct 17;8:788. doi: 10.3389/fphys.2017.00788. eCollection 2017. PMID 29089899
- [Background] Yow BG, Tennent DJ, Dowd TC, Loenneke JP, Owens JG. Blood Flow Restriction Training After Achilles Tendon Rupture. J Foot Ankle Surg. 2018 May-Jun;57(3):635-638. doi: 10.1053/j.jfas.2017.11.008. Epub 2018 Feb 21. PMID 29477554